CLINICAL TRIAL: NCT07203300
Title: BehavioRal Intervention Assisted by diGital Health Technology for Preventing Obesity Among Children（BRIGHT-POC）
Brief Title: Obesity Prevention in School-aged Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Collaborators: Shandong Maternal and Child Health Hospital (Unknown)
Responsible Party: Principal Investigator, Hai-Jun Wang, Professor in Department of Maternal and Child Health, School of Public Health, Peking University, Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NO.2025-072
Record Dates: First submitted 2025-09-24; First posted 2025-10-02 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Childhood Obesity Prevention
Keywords: Intervention; Obesity; Overweight; Children; School-aged
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Randomization will be performed after the baseline survey. The assessors measuring children's health indicators(e.g.,weight and height) will be blinded at follow up phases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A multi-level collaborative intervention (Experimental): The intervention includes: ① Health education: A trained teacher per class delivered 10 lessons during regular health classes, teaching five core messages in simple terms: not eating excessively; not drinking sugar--sweetened beverage; eating less high--energy food; less sedentary behaviours; performing more physical activity. ② Enhanced physical activity and BMI monitoring: physical education teachers guided daily moderate-to-vigorous activity. Teachers monthly measured height/weight, entered data into an app; children received feedback on BMI category and change. Weekly private weight measurements were also taken. ③ Family involvement: Implemented via offline meetings and a digital platform, the family-focused intervention provides health education and behavior change support, enabling parents to track BMI, log behaviors, review feedback, and access personalized consultations from medical professionals.
  Interventions: Behavioral: multicomponent, tiered intervention
- usual-care control (No Intervention): In the control group, participating school-aged children will receive no intervention during the study period and will continue their routine educational and management practices without modification. After the study is fully completed, control group school-aged children will have access to all intervention materials and health education resources developed for this project.

INTERVENTIONS:
Behavioral: multicomponent, tiered intervention — this intervention is a multi-level collaborative health management system-a digital health platform with four core modules: the Health Education Module, the Growth Monitoring Module, the Health Behavior Module, and the Home-School Partnership Module. The platform facilitates collaboration among schools, families, and hospitals as follows: Schools utilize the platform to manage tasks outlined in health policies, such as delivering educational content, monitoring student activity and diet, and recording monthly height/weight measurements via the Growth Monitoring Module.
  Families access the platform to receive multi-format health education, set goals, and review personalized feedback. The Home-School Partnership Module also enables communication for motivational interviewing sessions conducted by professionals offline or by phone.
  Hospitals leverage the platform to provide professional guidance and medical support, ensuring interventions are medically sound.
  Arms: A multi-level collaborative intervention

SUMMARY:
This cluster-randomized trial will develop and test an intervention technology for school-aged children. The program combines digital health technology and personalized behavior intervention through a WeChat platform.

Our main question is: Does this integrated approach improve obesity related outcomes and behaviors in children?

Investigator will:

* Compare children receiving the program with those receiving usual care.
* Track physical measures and health behaviors to measure effectiveness of intervention.
* Evaluate the program's safety, implementation process, and cost-effectiveness. Findings will determine if this approach should be expanded to more communities.

DETAILED DESCRIPTION:
This study is a one-year cluster randomized controlled trial (cRCT) to be conducted in 10 eligible primary schools. The schools will be randomly allocated to either the intervention group or the control group in a 1:1 ratio.

The technical core of this research involves the development of a multi-level collaborative health management technology system based on a WeChat platform. This platform will serve as the core intervention technology, providing functional support to the intervention group schools, their students, and parents.

Students in the control group schools will receive routine health education and physical examination procedures during the trial period.

To evaluate the effectiveness of this intervention technology, outcome measure data will be collected at multiple time points. All participating students will undergo physical measurements and health behavior questionnaire surveys at baseline (T0) and at the end of the intervention period (T1, i.e., 12 months post-baseline). The changes in primary and secondary outcome measures from baseline (T0) to the end of the intervention (T1) will be compared between the intervention and control groups.

Furthermore, to assess the long-term sustainability of the intervention effects, investigator plan to conduct follow-up surveys annually at 24 months (T2) and 36months (T3) post-intervention for both the intervention and control group students. Generalized linear mixed model or Generalized Estimating Equations (GEE) will be constructed to longitudinally analyze the differential trajectories of health outcomes between the two groups, thereby comprehensively evaluating the immediate effects and long-term sustainability of this integrated intervention technology.

ELIGIBILITY:
Inclusion Criteria:

* Schools will be selected based on the consent of primary leadership, demonstrated cooperation, and availability of necessary personnel (e.g., school health professionals). Classes will be limited to grades 2 and 3, with teachers showing strong willingness to collaborate. Both parental informed consent and child assent are required for participation.

Exclusion Criteria:

* Schools will be excluded if they cater to special populations (e.g., schools for children with disabilities), are involved in other obesity-related interventions within the specified timeframe, or plan to close or relocate within two years. Children will be excluded if they have histories of major organ diseases (e.g., cardiac, pulmonary, hepatic, or renal conditions), special diets (e.g., vegetarian), pathological eating disorders, physical limitations affecting activity, or obesity due to endocrine disorders or medication side effects.

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1400 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-10-09 (Estimated); Study Completion 2028-10-09 (Estimated)

PRIMARY OUTCOMES:
children's BMl change | at the end of the 12-month intervention
  Calculated based on height and weight using WHO standards. The primary outcome is the difference between two arms in the change of children's BMI from baseline to the end of the follow-up.

SECONDARY OUTCOMES:
Carotid Intima-Media Thickness,CIMT | at the end of the 12-month intervention
  Non-invasive measurement of carotid artery wall thickness via high-frequency ultrasound enables the assessment of subclinical atherosclerosis.
Body Mass Index Z-score(BMI-z) | at the end of the 12-month intervention; at 24-month follow-up; at 36-month follow-up
  The BMI-z score is calculated based on height and weight using WHO standards
Waist Circumference | at the end of the 12-month intervention; at 24-month follow-up; at 36-month follow-up
  Waist circumference is measured at the midpoint between the lower margin of the last palpable rib and the top of the iliac crest to evaluate central adiposity.
waist-to-Height Ratio, WHtR | at the end of the 12-month intervention; at 24-month follow-up; at 36-month follow-up.
  Calculated by dividing waist circumference by height, used as an indicator of fat distribution and risk for metabolic complications
Body Composition | at the end of the 12-month intervention; at 24-month follow-up; at 36-month follow-up
  Body fat percentage is assessed using a bioelectrical impedance analyzer (MC-780A, TANITA, Tokyo, Japan)
Children's Eating Behaviors | at the end of the 12-month intervention
  Assessed using the Children's Eating Behavior Questionnaire (CEBO), measuring dimensions such as food responsiveness satiety responsiveness, and emotional eating
Time Spent in Physical Activity | at the end of the 12-month intervention
  Evaluated using the Children's Leisure Activities Study Survey (CLAss), assessing the amount and type of physical activity and sedentary behavior, including screen time.
Pubertal Milestones Time | at the end of the 12-month intervention; at 24-month follow-up; at 36--month follow-up
  Pubertal milestones are defined as a sequence of observable, critical physiological markers that arise during the process of adolescent development. Typically assessed through self-report questionnaires, these milestones signify the individual's transition from childhood into sexual maturity.

IPD SHARING:
Plan to Share IPD: No
Individual participant data (lPD) will not be shared publicly due to ethical considerations. in accordance with the study's ethical approval and informed consent procedures, the data contain potentially sensitive personal health information and are protected to ensure participant confidentiality and privacy. Data access is therefore restricted to authorized research personnel only and cannot be made publicly available.